CLINICAL TRIAL: NCT04288908
Title: Trait Injustice and Its Effects on Anger Induced by Social Exclusion
Brief Title: Trait Injustice, Social Exclusion, and Anger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: InjusticeUJI
Record Dates: First submitted 2020-01-20; First posted 2020-02-28 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: General Population

STUDY DESIGN:
Intervention Model Description: The two conditions, based on the experimental task called Cyberball, will be: social inclusion and social exclusion.
Who Masked: Participant
Masking Description: Only participants will be masked to the assigned condition. The researcher has to be aware of the assigned condition to prepare the experimental task accordingly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social exclusion (Experimental): Cyberball is a ball-passing task in which the participant plays with two virtual players. In this condition, the user receives fewer passes than the other two participants (i.e., 10 out of 60).
  Interventions: Other: Cyberball experimental task
- Social inclusion (Active Comparator): Cyberball is a ball-passing task in which the participant plays with two virtual players. In this condition, the user receives a comparable number of passes than the other two participants (i.e., 20 out of 60).
  Interventions: Other: Cyberball experimental task

INTERVENTIONS:
Other: Cyberball experimental task — Cyberball is an experimental task in which participants have to pass a ball to two virtual players during 60 passes in total

SUMMARY:
Participants will be randomly allocated to one of two experimental conditions: social exclusion or social inclusion. Participants, but not experimenters will be blind to the assignment. Pre- and post-tests will be administered. Participants will be offered 7 euros in compensation for participating.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Signs the informed consent
* Can read and understand Spanish

Exclusion Criteria:

* Being younger than 18 years of age
* Does not sign the informed consent
* Cannot read or understand Spanish

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2020-02-08 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Change in Anger State from baseline to end of the experiment | The STAXI-2 will be administered twice: at Baseline and at the same day of Baseline assessment just after the experimental task (end of study)
  The STAXI-2 includes a measure of anger state (15 items) with responses ranging from 1="Absolutely not" to 3="A lot"
Trait Injustice | This measure will be administered at Baseline
  The Trait Injustice Experiences Questionnaire is a measure of perceived trait injustice beliefs that has 12 items, with responses ranging from 0="never" to 4="always". This measure will be used as moderator of the effects of the experiment on anger

SECONDARY OUTCOMES:
Frustration Discomfort Scale | This measure will be administered at Baseline
  This is a measure of frustration intolerance. The scale has 28 items that are gouped in 4 subscales. Items have a 1-to-5 response scale ranging from "nothing" to "a lot". In addition to trait injustice, this measure will also be used in secondary analyses as a moderator of the effects of the experiment on anger
Change in State Injustice from baseline to end of the experiment | This measure will be administered twice: at Baseline and at the same day of Baseline assessment just after the experimental task (end of study)
  The State Injustice Experiences Questionnaire is a measure of perceived state injustice beliefs that has 12 items, with responses ranging from 0="never" to 4="always". This measure will be used as an experimental check (whether exclusion in the experiment effectively increased the sense of injustice in the short term)
Change in State Anxiety from baseline to end of the experiment | This measure will be administered twice: at Baseline and at the same day of Baseline assessment just after the experimental task (end of study)
  The STAI-S is a measure of perceived state anxiety that has 20 items, with responses ranging from 0="not at all" to 3="a lot". This measure will be used as an experimental check (whether exclusion in the experiment effectively increased anxiety in the short term)
Cyberball Experiences post-experimental check Questionnaire | This measure will be administered at the same day of Baseline assessment just after the experimental task (end of study)
  In addition to exploring the effects of the experimental task on anxiety and anger, the Cyberball includes a measure of impact of the task on perceived inclusion and related concepts (isolation, belonging, perceived number of passes received, etc.). This will also be used as an experimental check

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Psycholoy. Jaume I University, Castellon, Spain

IPD SHARING:
Plan to Share IPD: No
Only the main PI will have access to the data.